CLINICAL TRIAL: NCT05674565
Title: The Neuroprotective Impact of Magnesium Sulphate Therapy for Preterm Deliveries. Loading Dose Alone Strategy Versus Loading Plus Maintenance Dose Strategy.
Brief Title: Magnesium Sulphate Neuroprotective Strategies for Preterm Deliveries
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Hytham Atia, Associate professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MGSULPH NEUROPROTECT EGYPT
Record Dates: First submitted 2022-11-19; First posted 2023-01-06 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Premature Birth; NEUROPROTECTION; MAGNESIUM SULPHATE; Cerebral Palsy; Neonatal Death
Keywords: CEREBRAL PALSY; PRETERM BIRTH; NEUROPROTECTION; NEONATAL DEATH; MAGNESIUM SULPHATE
MeSH Terms: conditions — Premature Birth; Cerebral Palsy; Perinatal Death | interventions — Short-Wave Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Loading dose only (Experimental): Those receiving only the loading dose of magnesium sulphate 4 gm infusion over 20 minutes therapy within one hour before delivery without the maintenance dose
  Interventions: Drug: Magnesium sulfate loading dose only
- Loading plus maintenance dose (Experimental): Receiving magnesium sulphate loading 4 gm infusion over 20 minutes, followed by maintenance therapy 1gm per hour infusion until delivery or completion of 24 hours, the sooner.
  Interventions: Drug: Magnesium sulfate loading with maintenance dose
- Control (No Intervention): comparable number of women who did not receive magnesium sulphate neuroprotection for any reason

INTERVENTIONS:
Drug: Magnesium sulfate loading with maintenance dose — 4 gm MgSo4 loading over 20 minutes followed by 1 gm per hour maintenance till delivery
  Other Names: complete therapy
  Arms: Loading plus maintenance dose
Drug: Magnesium sulfate loading dose only — 4 gm MgSo4 loading over 20 minutes within one hour before delivery
  Other Names: short therapy
  Arms: Loading dose only

SUMMARY:
A Cochrane systematic review has confirmed that fetal exposure to magnesium sulphate given before preterm birth has a neuroprotective role. This review also showed a significant reduction in the rate of gross motor dysfunction in early childhood. Early Preterm birth (< 34+0 weeks) and very low birthweight (< 1,500 g) are the principal risk factors for cerebral palsy. Multiple pregnancy accounts for over 10% of preterm births and has a higher incidence of cerebral palsy than singleton pregnancy (twins have 7 times and triplets 47 times the risk of cerebral palsy compared with singletons).

DETAILED DESCRIPTION:
Many of these patients come or get diagnosed as eminent preterm delivery very soon before the real delivery happens and are not able to complete the recommended therapy of loading and maintenance strategy for at least complete 4 hours before delivery.

Till now, there is a gap and lack of knowledge regarding the value of loading dose only as sufficient and effective strategy for neuroprotection compared to full therapy, which needs more health costs, longer monitoring and carries more risk for the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Women at risk of preterm birth who are between 24+0 and 33+6 weeks of gestation.
2. When early preterm birth is planned or expected within 24 h, regardless of:

   * Plurality or parity
   * Reason for the risks of preterm birth
   * Anticipated mode of birth
   * Whether antenatal corticosteroids have been given or not

Exclusion Criteria:

* Women with known Hypersensitivity to magnesium
* Caution regarding dosage for patients with renal impairment
* Preterm delivery after 34 weeks

Ages: 24 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 336 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Neonatal Neurological insult | at 18 months age after delivery
  The incidence of neurological insults during the first year of life (including cerebral palsy, brain leukomalacia, intraventricular hemorrhage, and neonatal seizures)
Maternal toxicity | from start of therapy, till 12 hours after end of therapy
  Risk of maternal magnesium sulphate toxicity (affected reflexes, respiratory and cardiac), postpartum hemorrhage.
Postpartum hemorrhage | first 24 hours after delivery
  Risk of primary postpartum hemorrhage

SECONDARY OUTCOMES:
Late appearing neurologic insults | at 24 months age after delivery
  Risk of gross motor delay, epilepsy, impaired fine motor skills, sensorineural (hearing and vision) impairment, and possibly two years of age developmental quotient.
Neonatal death | 28 days from birth
  Death within first 28 days after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Hytham Atia, M.D., Study Chair — Zagazig University; Amro Alnemr, M.D., Principal Investigator — Zagazig University; Mohamed Lashin, M.D., Principal Investigator — Zagazig University; Sherief M El Gebaly, M.D., Principal Investigator — Zagazig University; Mohamed Arafa, M.D., Principal Investigator — Zagazig University
Locations (1):
- Faculty of medicine, Zagazig University, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shennan A, Suff N, Jacobsson B, Simpson JL, Norman J, Grobman WA, Bianchi A, Mujanja S, Valencia CM, Mol BW. FIGO good practice recommendations on magnesium sulfate administration for preterm fetal neuroprotection. Int J Gynecol Obstet. 2021;155(1):31-33. doi:10.1002/ijgo.13856.
- [Background] Usman S, Foo L, Tay J, Bennett PR, Lees C. Use of magnesium sulfate in preterm deliveries for neuroprotection of the neonate. Obstet Gynaecol. 2017;19(1):21-28. doi:10.1111/tog.12328